CLINICAL TRIAL: NCT03363386
Title: Effects oF Resistive Exercise or Proprioceptive Exercise Training on Balance and Superficial Sense of Patients With Type 2 Diabetes Mellitus
Brief Title: Effects Of Resistive Exercise or Proprioceptive Exercise Training Among Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Yeditepe U
Record Dates: First submitted 2017-11-10; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: aerobic exercise; dynamic balance; functional capacity; HbA1c; proprioceptive exercise training
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The sample of study consists of patients with Type 2 Diabetes Mellitus (DM) got diagnosed at least 6 months and who referred to Fitness Center in Pendik Arif Nihat Asya Kültür Merkezi Istanbul Turkey by a medical doctor between December 2016- March 2017. The study included in 30 patients (24F, 6M) with T2DM. The patients who met inclusion criteria are divided into two groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive Exercise Group (PG) (Experimental): Aerobic Exercise Proprioceptive Exercises
  Interventions: Procedure: Proprioceptive Exercises; Procedure: Aerobic Exercise
- Resistive Exercise Group (RG) (Active Comparator): Aerobic Exercise Resistive Exercises
  Interventions: Procedure: Resistive Exercises; Procedure: Aerobic Exercise

INTERVENTIONS:
Procedure: Proprioceptive Exercises — Patients trained for proprioceptive exercises
  Arms: Proprioceptive Exercise Group (PG)
Procedure: Resistive Exercises — Patients trained for resistive exercises
  Arms: Resistive Exercise Group (RG)
Procedure: Aerobic Exercise — Patients were educated with treadmill walking for 30 minutes of each exercise session

SUMMARY:
The aim of the study is to investigate proprioceptive exercises training combined with aerobic exercises and resistive exercises training combined with aerobic exercises on dynamic balance and superficial sense. The patients were randomly divided into Proprioceptive Exercise Training Group (PG) (n=15) and Resistive Exercise Training Group (RG) (n=15). All subjects were included exercise education program and both groups had trained aerobic exercise program for walking on treadmill (2times/wk. 6 week duration).

DETAILED DESCRIPTION:
The aim of the study is to investigate proprioceptive exercises training combined with aerobic exercises and resistive exercises training combined with aerobic exercises on dynamic balance and superficial sense. The study included 30 volunteers with Type 2 Diabetes Mellitus(T2DM) who were referred to Fitness Center Arif Nihat Asya Kültür Merkezi Istanbul, Turkey by a medical doctor between December 2016- March 2017 and got diagnosed and followed up at least 6 month before. Glycemic control of all the participants were assessed according to fasting blood glucose and glycolated hemoglobin (HbA1c). Waist and hip circumference was recorded in centimeters. Six minute walking test (6MWT) was used to determine functional capacity of participants. We evaluated the dynamic balance of patients by Prokin PK200, Italy. Five parameters were obtained from Prokin as; Perimeter Length (PL), Area gap percentade (AGP) Medium Speed (MS), Anteroposterior equilibrium (AP) and Mediolateral equilibrium (ML). Proprioception assessment was done with angle reproduction test in direction of dorsiflexion and plantar flexion and deviations were recorded. Superficial sense was assessed with two point discrimination test and vibration threshold was evaluated by biothesiometer. Lower extremity muscles strength were assessed with handheld dynamometer (PowerTrack II commander, JTech Medical, Midvale, UT). The patients were randomly divided into Proprioceptive Exercise Training Group (PG) and Resistive Exercise Training Group (RG). All subjects were included exercise education program and both groups had trained aerobic exercise program for walking on treadmill (2times/wk. 6 week duration). The proprioceptive exercise program was applied in PG and the resistive exercise program was applied in RG twice a week and for duration 6 week.

ELIGIBILITY:
Inclusion Criteria:

* Participating to the study in a voluntary basis
* Patients with 30-60 years old
* Getting diagnosed with Type 2 Diabetes Mellitus (DM) at least 6 months.

Exclusion Criteria:

* Unstable cardiac condition
* Uncontrolled Diabetes Mellitus
* Uncontrolled Hypertension
* Symptomatic Heart Failure, unstable angina
* Peripheral Arterial Occlusive Disease
* Diabetic foot ulcers
* Part/total foot amputation
* Myocardial infarction within 3 months prior to study
* Coronary Artery Bypass within 3 months prior to study
* Cerebrovascular ischemia/stroke (including TIA) within 3 months of study
* Severe retinopathy, nephropathy
* Thyroid Dysfunctions (hyperthyroidism, hypothyroidism).

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c level | 6 weeks
  It was evaluated for metabolic control with patient's routine controls in their clinics follow-up. At the end of the study, this metabolic variable was evaluated again in order to observe changes
Waist and Hip Circumferences | 6 weeks
  It represents risks for cardiovascular diseases.
Six minute walking test | 6 weeks
  Functional capacity of the patients was evaluated through 6 minute walking test
Dynamic balance assessment | 6 weeks
  Prokin PK 200 was used for dynamic balance assessment
Vibration Perception Threshold Assessment | 6 weeks
  Biothesiometer was used for determining vibration perception threshold
Lower Extremity Muscle Strength | 6 weeks
  Commander myometer was used for muscle strength assessment
Proprioception Assesment | 6 weeks
  Angle reproduction test was used
Two Point Discrimination Test | 6 weeks
  aesthesiometer was used to determine two point discrimination sensation
Change in fasting blood glucose level | 6 weeks
  It was evaluated for metabolic control with patient's routine controls in their clinics follow-up. At the end of the study, this metabolic variable was evaluated again in order to observe changes

CONTACTS AND LOCATIONS:
Overall Officials: Guzin Kaya Aytutuldu, M.Sc., Principal Investigator — Yeditepe University, Health Sciences Faculty, Department of Physiotherapy and Rehabilitation; Feryal Subasi, Professor, Study Chair — Yeditepe University, Health Sciences Faculty, Department of Physiotherapy and Rehabilitation; Gülgün Arslan, MD, Study Chair — Istanbul Pendik Kaynarca Outpatient Policlinic Diabetes Center; Elif Develi, M.Sc., Study Chair — Yeditepe University, Health Sciences Faculty, Department of Physiotherapy and Rehabilitation

IPD SHARING:
Plan to Share IPD: No